CLINICAL TRIAL: NCT05153863
Title: Performance and Safety of the C Scope Visualization System in Arthroscopic Procedures - A Prospective Study
Brief Title: C Scope Visualization System Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIT Ortho (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZSC-DVER-330-02-PR32
Record Dates: First submitted 2021-11-30; First posted 2021-12-10 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Knee Injuries and Disorders; Shoulder Disease; Shoulder Injuries
Keywords: Visualization; Illumination; Arthroscopic Procedures
MeSH Terms: conditions — Knee Injuries; Disease; Shoulder Injuries

STUDY DESIGN:
Intervention Model Description: Evaluation of the performance and safety of the C Scope Visualization System in the illumination and visualization of joints during diagnostic procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm C-Scope Visualization System (Experimental): The C Scope Visualization System is indicated to be used by a trained physician to provide illumination and visualization in arthroscopic procedures of an interior cavity of the body through a surgical opening.
  Interventions: Device: C Scope Visualization System

INTERVENTIONS:
Device: C Scope Visualization System — The C Scope Visualization System is indicated to be used by a trained physician to provide illumination and visualization in arthroscopic procedures of an interior cavity of the body through a surgical opening.

SUMMARY:
Evaluation of the performance and safety of the C Scope Visualization System

DETAILED DESCRIPTION:
The C Scope Visualization System Prospective Study is a post-market, single-arm, prospective, multicenter study conducted in the United States.

The purpose of the study is to evaluate the performance and safety of the C Scope Visualization System in the illumination and visualization of joints from diagnostic procedure through 1-week and 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject can fluently speak and read English
* Subject is able to provide informed consent
* Subject agrees to all protocol-required follow-ups
* Subject meets the C Scope Indications for Use according to approved labeling

Exclusion Criteria:

* History of open surgery to the index joint resulting in scarring that might inhibit evaluation with the C Scope Visualization System
* Suspected fracture of joint structures
* Subject has any contraindications listed in the approved labeling including active infection
* In the opinion of the investigator, it is not in the subject's best interest to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Physician-rated procedural (diagnostic only) illumination and visualization with the C-Scope Visualization System | Peri procedure
  Physician-rated procedural (diagnostic only) illumination and visualization of the areas with the C-Scope Visualization System of the joint intended to be evaluated using a 5-point scale:

SECONDARY OUTCOMES:
Physician-rated confidence of diagnosis with the C-Scope Visualization System | Peri procedure
  Physician-rated confidence of diagnosis following needle arthroscopy attributed to visualization performance of the device using a 5-point scale
Physician-rated needle arthroscopy procedural ease with the C-Scope Visualization System | Peri procedure
  Physician-rated needle arthroscopy procedural ease using a 5- point scale
Procedure time with the C-Scope Visualization System | Peri procedure
  Procedure time (from start of arthroscopy to end of procedure)

OTHER OUTCOMES:
Safety Adverse Events | 1 week and 1 month post procedure
  Adverse events/serious adverse event rates related to the procedure or device

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Hanson, MD, Principal Investigator — Desert Orthopaedic Center
Locations (1):
- Desert Orthopaedic Center, Henderson, Nevada, United States

IPD SHARING:
Plan to Share IPD: No